CLINICAL TRIAL: NCT02954991
Title: A Parallel Phase 2 Study of Glesatinib, Sitravatinib or Mocetinostat in Combination With Nivolumab in Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Phase 2 Study of Glesatinib, Sitravatinib or Mocetinostat in Combination With Nivolumab in Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated as a result of Sponsor portfolio reprioritization.
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRTX-500
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — glesatinib; sitravatinib; mocetinostat; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glesatinib and Nivolumab (Experimental): Glesatinib oral tablet administered twice daily in combination with Nivolumab administered as 240 mg IV every 2 weeks or 480 mg IV every 4 week
  Interventions: Drug: Glesatinib; Drug: Nivolumab
- Sitravatinib and Nivolumab (Experimental): Sitravatinib oral capsule administered daily in combination with nivolumab administered as 240 mg IV every 2 weeks or 480 mg IV every 4 week
  Interventions: Drug: Sitravatinib; Drug: Nivolumab
- Mocetinostat and Nivolumab (Experimental): Mocetinostat oral capsule administered three times weekly in combination with nivolumab administered as 240 mg IV every 2 weeks or 480 mg IV every 4 week
  Interventions: Drug: Mocetinostat; Drug: Nivolumab

INTERVENTIONS:
Drug: Glesatinib — Glesatinib is a small molecule multi-targeted receptor tyrosine kinase inhibitor
  Other Names: MGCD265
  Arms: Glesatinib and Nivolumab
Drug: Sitravatinib — Sitravatinib is a small molecule inhibitor of receptor tyrosine kinases.
  Other Names: MGCD516
  Arms: Sitravatinib and Nivolumab
Drug: Mocetinostat — Mocetinostat is an HDAC inhibitor.
  Other Names: MGCD01013
  Arms: Mocetinostat and Nivolumab
Drug: Nivolumab — nivolumab is a programmed death receptor-1 (PD-1) blocking antibody
  Other Names: Opdivo

SUMMARY:
The study will evaluate the clinical activity of nivolumab in combination with 3 separate investigational agents, glesatinib, sitravatinib, or mocetinostat.

DETAILED DESCRIPTION:
Glesatinib is an orally administered multi-targeted tyrosine kinase inhibitor (TKI) that primarily targets the Axl and Mesenchymal-Epithelial Transition (MET) receptors. Sitravatinib is an orally-available, potent small molecule inhibitor of a closely related spectrum of receptor tyrosine kinases (RTKs) including MET, Axl, MERTK, VEGFR family, PDGFR family, KIT, FLT3, Trk family, RET, DDR2 and selected Eph family members. Mocetinostat is an orally administered histone deacetylase (HDAC) inhibitor. Nivolumab is a human IgG monoclonal antibody that binds to the programmed cell death-1(PD-1) receptor and blocks its interaction with programmed cell death ligand-1 (PD-L1) and PD-L2, releasing PD-1 pathway-mediated inhibition of the immune response including anti-tumor immune response. Combining an immunotherapeutic PD-L1 checkpoint inhibitor with an agent that has both immune modulatory and antitumor properties could enhance the antitumor efficacy observed with either agent alone.

The study will begin with a lead-in dose escalation evaluation of two dose levels of each investigational agent in combination with nivolumab. Following completion of the lead-in dose escalation, enrollment into the Phase 2 study will proceed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-small cell lung cancer.
* Prior treatment with a checkpoint inhibitor (as appropriate per cohort)
* Adequate bone marrow and organ function

Exclusion Criteria:

* Uncontrolled tumor in the brain
* Unacceptable toxicity with prior checkpoint inhibitor
* Impaired heart function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Yuma Regional Medical Center, Yuma, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego, La Jolla, California
  - University of California San Francisco Comprehensive Cancer Center, San Francisco, California
  - University of California Los Angeles - Torrance - Community Cancer Care, Santa Clarita, California
  - Rocky Mountain Cancer Centers - Denver - Midtown, Denver, Colorado
  - Baptist Health, Louisville, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Oncology Hematology Care-Blue Ash, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Hematology Oncology Associates - Barnett Office, Medford, Oregon
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Texas Oncology - South Austin, Austin, Texas
  - USOR - Texas Oncology - Denison Cancer Center, Denison, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Cancer Specialist, Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across 25 sites in the United States from November 2016 to November 2021.
Pre-assignment Details: Participants enrolled: 161, 156 included for sitravatinib + nivolumab and 5 for glesatinib + nivolumab. Main study groups: CIT Experienced and CIT Naive. Enrollment into glesatinib cohorts was discontinued November 2017. Enrollment into mocetinostat cohorts was never initiated. These decisions were not based on participant safety in Study MRTX-500.
Groups:
- CIT Experienced: Sitravatinib and Nivolumab: Participants who had previously received checkpoint inhibitor therapy (CIT) received sitravatinib 120 mg oral capsules once daily (QD) in combination with nivolumab 240 mg every 2 weeks or 480 mg every 4 weeks intravenously.
- CIT Naïve: Sitravatinib and Nivolumab: Participants who had not previously received CIT received sitravatinib 120 mg oral capsules QD in combination with nivolumab 240 mg every 2 weeks or 480 mg every 4 weeks intravenously.
- Glesatinib and Nivolumab: Participants received glesatinib 500 mg oral tablets twice daily in combination with nivolumab 240 mg every 2 weeks intravenously.
Period: Overall Study
Arm/Group | CIT Experienced: Sitravatinib and Nivolumab | CIT Naïve: Sitravatinib and Nivolumab | Glesatinib and Nivolumab
Started | 124 | 32 | 5
Received Any Study Treatment | 124 | 32 | 5
Completed | 0 | 0 | 0
Not Completed | 124 | 32 | 5
Not completed — Death | 92 | 11 | 2
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Withdrawal by Subject | 9 | 8 | 1
Not completed — Study Terminated by Sponsor | 18 | 10 | 1
Not completed — Miscellaneous | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population was defined as all participants who received at least 1 dose of any study treatment (sitravatinib, glesatinib, or nivolumab). 1 participant has been excluded from the analysis as the PD-L1 status could not be confirmed due to a missing laboratory sample.
Groups:
- Glesatinib and Nivolumab: Participants received glesatinib 500 mg oral tablets twice daily in combination with nivolumab 240 mg every 2 weeks or 480 mg every 4 weeks intravenously.
- Total: Total of all reporting groups
Arm/Group | CIT Experienced: Sitravatinib and Nivolumab | CIT Naïve: Sitravatinib and Nivolumab | Glesatinib and Nivolumab | Total
Number analyzed (Participants) | 124 | 32 | 5 | 161
Age, Customized [Count of Participants; unit: Participants] — The data collected for this study only supports age customized as a baseline measure. Age was summarized as a continuous outcome, no age was specified in the statistical analysis plan.
  Participants
    30 to 89 years | 124 | 32 | 5 | 161
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 20 | 2 | 88
  Male | 58 | 12 | 3 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 0 | 7
  Not Hispanic or Latino | 118 | 29 | 5 | 152
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  [Not specified]: American Indian or Alaska Native | 1 | 0 | 0 | 1
  [Not specified]: Asian | 3 | 1 | 0 | 4
  [Not specified]: Native Hawaiin or Other Pacific Islander | 0 | 1 | 0 | 1
  [Not specified]: Black or African American | 8 | 3 | 2 | 13
  [Not specified]: White | 107 | 26 | 3 | 136
  [Not specified]: Other | 5 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Description: ORR is defined as the percentage of participants that were documented to have a confirmed complete response (CR) or partial response (PR) as defined by RECIST v1.1.
Time Frame: Up to 40.6 months
Population: The Full Analysis Set (FAS) was defined as all participants who received at least 1 dose of both study treatments (sitravatinib or glesatinib) and nivolumab. Data was only planned to be reported for participants in the Phase 2 study, so no data is present for the 5 participants who received glesatinib in the lead- in phase only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CIT Experienced: Sitravatinib and Nivolumab | CIT Naïve: Sitravatinib and Nivolumab
Number analyzed (Participants) | 124 | 32
percentage of participants | 15.3 [9.5 to 22.9] | 25 [11.5 to 43.4]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any event that first occur or increase in severity on or after the first dose of study treatment and not more than 28 days after the last dose of study treatment and prior to the initiation of subsequent systemic anti- cancer therapy.
  Any clinically significant changes in laboratory tests were recorded as TEAEs.
Time Frame: Day 1 up to 28 days after the last dose (median time on treatment was: CIT experienced 3.7 months; CIT naïve 4.8 months)
Population: The Safety Population was defined as all participants who received at least 1 dose of any study treatment (sitravatinib, glesatinib, or nivolumab). Per statistical analysis plan, only AEs for sitravatinib + nivolumab will be summarized. TEAE tables for glesatinib + nivolumab were not produced and therefore will not be reported here.
Measure: Count of Participants; unit: Participants
Arm/Group | CIT Experienced: Sitravatinib and Nivolumab | CIT Naïve: Sitravatinib and Nivolumab
Number analyzed (Participants) | 124 | 32
Participants | 123 | 32

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time in months from date of the first documentation of objective response (CR or PR) to the first documentation of objective progressive disease (PD) or to death due to any cause in the absence of documented PD. (Be aware, the population analyzed here is the Clinical Activity Evaluable Population and not the Full Analysis Set as used in outcome measure 1).
Time Frame: Up to 38.8 months
Population: Clinical Activity Evaluable Population was defined as all participants who received at least 1 dose of both study treatments (sitravatinib or glesatinib) and nivolumab, had an evaluable baseline tumor assessment, and ≥ 1 postbaseline tumor assessment. DOR was only calculated for the participants that achieved a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CIT Experienced: Sitravatinib and Nivolumab | CIT Naïve: Sitravatinib and Nivolumab
Number analyzed (Participants) | 19 | 8
months | 11.0 [3.7 to 13.1] | 11.1 [3.7 to NA] — Insufficient number of participants with events

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first dose of study drug to the date of PD or death due to any cause in the absence of documented PD, whichever occurs first.
Time Frame: Up to 40.6 months
Population: The FAS was defined as all participants who received at least 1 dose of both study treatment (sitravatinib or glesatinib) and nivolumab. Data was only planned to be collected for participants in the Phase 2 study, so no data is present for the 5 participants who received glesatinib in the lead-in phase only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CIT Experienced: Sitravatinib and Nivolumab | CIT Naïve: Sitravatinib and Nivolumab
Number analyzed (Participants) | 124 | 32
months | 5.4 [4.2 to 5.7] | 7.1 [4.0 to 13.1]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of study drug to the date of death due to any cause.
Time Frame: Up to 43.8 months
Population: FAS was defined as all participants who received at least 1 dose of both study treatments (sitravatinib or glesatinib) and nivolumab. Data was only planned to be collected for participants in the Phase 2 study, so no data is present for the 5 participants who received glesatinib in the lead-in phase only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CIT Experienced: Sitravatinib and Nivolumab | CIT Naïve: Sitravatinib and Nivolumab
Number analyzed (Participants) | 124 | 32
months | 11.5 [8.7 to 15.0] | NA [9.8 to NA] — The overall median value for CIT naive was not reached, and the upper limit of confidence interval was not estimable. Only 11 events and 21 patients censored, therefore not enough data to estimate the median survival and upper limit of 95% CI.

6. Secondary Outcome: Blood Plasma Concentrations
Description: Predose (trough) concentrations for sitravatinib
Time Frame: Cycle 1 Day 1 through Cycle 5 Day 1
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Cycle 1 Day 15: Summary of all patients sitravatinib 120mg QD trough concentrations at C1D15
- Cycle 2 Day 1: Summary of all patients sitravatinib 120mg QD trough concentrations at C2D1
- Cycle 2 Day 15: Summary of all patients sitravatinib 120mg QD trough concentrations at C2D15
- Cycle 3 Day 1: Summary of all patients sitravatinib 120mg QD trough concentrations at C3D1
- Cycle 5 Day 1: Summary of all patients sitravatinib 120mg QD trough concentrations at C5D1
Arm/Group | Cycle 1 Day 15 | Cycle 2 Day 1 | Cycle 2 Day 15 | Cycle 3 Day 1 | Cycle 5 Day 1
Number analyzed (Participants) | 117 | 82 | 57 | 39 | 11
ng/ml | 76.57 (51.041) | 59.25 (36.759) | 52.87 (26.265) | 46.41 (26.183) | 30.04 (12.239)

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after the last dose
Description: Participants were assessed for all-cause mortality from their first dose to study completion (up to approximately 46 months). SAEs and Other AEs were assessed from first dose to 28 days following last dose (up to approximately 46 months + 28 days).
Groups:
- CIT Experienced: Sitravatinib and Nivolumab: Participants who had previously experienced checkpoint inhibitor therapy (CIT) received sitravatinib 120 mg oral capsules once daily (QD) in combination with nivolumab 240 mg every 2 weeks or 480 mg every 4 weeks intravenously.
- CIT Naive: Sitravatinib and Nivolumab: Participants who had not previously experienced CIT received sitravatinib 120 mg oral capsules QD in combination with nivolumab 240 mg every 2 weeks or 480 mg every 4 weeks intravenously.
Arm/Group | CIT Experienced: Sitravatinib and Nivolumab | CIT Naive: Sitravatinib and Nivolumab | Glesatinib and Nivolumab
All-Cause Mortality (participants affected / at risk) | 92/124 | 11/32 | 2/5
Serious Adverse Events (participants affected / at risk) | 62/124 | 17/32 | 1/5
Other Adverse Events (participants affected / at risk) | 122/124 | 31/32 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIT Experienced: Sitravatinib and Nivolumab (N=124) | CIT Naive: Sitravatinib and Nivolumab (N=32) | Glesatinib and Nivolumab (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 3 (3) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIT Experienced: Sitravatinib and Nivolumab (N=124) | CIT Naive: Sitravatinib and Nivolumab (N=32) | Glesatinib and Nivolumab (N=5)
Anaemia (Blood and lymphatic system disorders) | 27 (27) | 11 (11) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 12 (12) | 4 (4) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 5 (5) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 30 (30) | 13 (13) | 0 (0)
Vision blurred (Eye disorders) | 6 (6) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 8 (8) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 23 (23) | 5 (5) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 31 (31) | 12 (12) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 79 (79) | 20 (20) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 17 (17) | 5 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 9 (9) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 8 (8) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 (13) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 62 (62) | 16 (16) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 20 (20) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 48 (48) | 12 (12) | 1 (1)
Asthenia (General disorders) | 8 (8) | 3 (3) | 0 (0)
Chills (General disorders) | 7 (7) | 2 (2) | 0 (0)
Fatigue (General disorders) | 77 (77) | 21 (21) | 2 (2)
Gait disturbance (General disorders) | 7 (7) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 12 (12) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 11 (11) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 17 (17) | 8 (8) | 1 (1)
Pyrexia (General disorders) | 15 (15) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 12 (12) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 4 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 15 (15) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 28 (28) | 4 (4) | 2 (2)
Amylase increased (Investigations) | 9 (9) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 27 (27) | 8 (8) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 18 (18) | 4 (4) | 0 (0)
Blood creatinine increased (Investigations) | 9 (9) | 4 (4) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 5 (5) | 6 (6) | 0 (0)
Lipase increased (Investigations) | 14 (14) | 4 (4) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (11) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 15 (15) | 5 (5) | 0 (0)
Weight decreased (Investigations) | 57 (57) | 13 (13) | 0 (0)
White blood cell count decreased (Investigations) | 6 (6) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 62 (62) | 19 (19) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 26 (26) | 8 (8) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 7 (7) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 11 (11) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 33 (33) | 8 (8) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 16 (16) | 7 (7) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (7) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (23) | 6 (6) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 25 (25) | 8 (8) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 31 (31) | 10 (10) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (20) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (21) | 5 (5) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 13 (13) | 8 (8) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (12) | 7 (7) | 1 (1)
Dizziness (Nervous system disorders) | 19 (19) | 7 (7) | 0 (0)
Dysgeusia (Nervous system disorders) | 14 (14) | 7 (7) | 0 (0)
Headache (Nervous system disorders) | 18 (18) | 6 (6) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 10 (10) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 7 (7) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 15 (15) | 7 (7) | 0 (0)
Proteinuria (Renal and urinary disorders) | 14 (14) | 7 (7) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (32) | 15 (15) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 42 (42) | 10 (10) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (30) | 10 (10) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 20 (20) | 8 (8) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 13 (13) | 6 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (13) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 41 (41) | 11 (11) | 0 (0)
Hypotension (Vascular disorders) | 8 (8) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment into glesatinib cohorts was discontinued in November 2017 as a result of Sponsor portfolio reprioritization. The analysis and reporting of this treatment arm is limited and will be summarized for selected tables only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT02954991/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT02954991/SAP_001.pdf
  • Informed Consent Form (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT02954991/ICF_002.pdf